CLINICAL TRIAL: NCT04961112
Title: Evaluating the Efficacy of Cranial Electrotherapy Stimulation in Mitigating Anxiety-induced Cognitive Deficits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Nathan Ward, Associate Professor, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1908026
Record Dates: First submitted 2021-07-01; First posted 2021-07-14 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Cognitive Deficit
Keywords: Cranial electrotherapy stimulation; Executive functioning; Induced Anxiety; Cognition; Threat of shock; Heart rate variability
MeSH Terms: conditions — Anxiety Disorders; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All study staff are blinded to active and sham brain stimulation devices until the completion of data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental - Induced Anxiety (Experimental): Participants will be administered a shock procedure in which they are exposed to safe electrical shock that will be gradually increase from (1) 30 milliseconds to (4) 80 milliseconds to an individual threshold that is uncomfortable but not painful. Participants will be told they may receive additional shocks for poor performance during cognitive assessments.
  Participants will be administered cranial electrotherapy stimulation with a frequency of .5 Hz and a current of 100 microamps during 30 minutes of cognitive assessments of task switching, inhibition (stroop), working memory (n-back), and processing speed (simple reaction time).
  Interventions: Device: Cranial Electrotherapy Stimulation
- Experimental - No Induced Anxiety (Experimental): Participants will be administered a shock procedure in which they are exposed to safe electrical shock that will be gradually increase from (1) 30 milliseconds to (4) 80 milliseconds to an individual threshold that is uncomfortable but not painful. After this procedure, the shock belt will be turned off. Participants will be told they will not receive additional shocks during cognitive assessments.
  Participants will be administered cranial electrotherapy stimulation with a frequency of .5 Hz and a current of 100 microamps during 30 minutes of cognitive assessments of task switching, inhibition (stroop), working memory (n-back), and processing speed (simple reaction time).
  Interventions: Device: Cranial Electrotherapy Stimulation
- Sham - Induced Anxiety (Sham Comparator): Participants will be administered a shock procedure in which they are exposed to safe electrical shock that will be gradually increase from (1) 30 milliseconds to (4) 80 milliseconds to an individual threshold that is uncomfortable but not painful. Participants will be told they may receive additional shocks for poor performance during cognitive assessments.
  Participants will be administered sham cranial electrotherapy stimulation with no current during 30 minutes of cognitive assessments of task switching, inhibition (stroop), working memory (n-back), and processing speed (simple reaction time).
  Interventions: Device: Sham Cranial Electrotherapy Stimulation
- Sham - No Induced Anxiety (Sham Comparator): Participants will be administered a shock procedure in which they are exposed to safe electrical shock that will be gradually increase from (1) 30 milliseconds to (4) 80 milliseconds to an individual threshold that is uncomfortable but not painful. After this procedure, the shock belt will be turned off. Participants will be told they will not receive additional shocks during cognitive assessments.
  Participants will be administered sham cranial electrotherapy stimulation with no current during 30 minutes of cognitive assessments of task switching, inhibition (stroop), working memory (n-back), and processing speed (simple reaction time).
  Interventions: Device: Sham Cranial Electrotherapy Stimulation

INTERVENTIONS:
Device: Cranial Electrotherapy Stimulation — Participants will receive cranial electrotherapy stimulation stimulation on one of two separate visits (within-subjects).
  Other Names: Transcranial Pulsed Current Stimulation; Cranial Electrical Stimulation
  Arms: Experimental - Induced Anxiety; Experimental - No Induced Anxiety
Device: Sham Cranial Electrotherapy Stimulation — Participants will receive sham stimulation on one of two separate visits (within-subjects).
  Arms: Sham - Induced Anxiety; Sham - No Induced Anxiety

SUMMARY:
This study investigates the potential of cranial electrotherapy stimulation to mitigate anxiety induced cognitive deficits

ELIGIBILITY:
Inclusion Criteria:

* Between 18-28 years old

Exclusion Criteria:

* History of diagnosis with a neurological or psychiatric disorder.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Task switching | 68 weeks
  Switch cost (mean switch reaction time- mean stay reaction time)
Working memory (N-back) | 68 weeks
  2-back condition mean accuracy
Inhibition (Stroop) | 68 weeks
  Stroop interference cost (mean incongruent reaction time- mean congruent reaction time)
Processing speed (Simple reaction time task) | 68 weeks
  Mean reaction time

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Medford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No